CLINICAL TRIAL: NCT01954875
Title: Establishment of a Human Tissue Bank for Studying the Microbial Etiology of Neurodegenerative Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Study no longer funded
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CHS-Neurology-ALS stool sample
Record Dates: First submitted 2013-03-30; First posted 2013-10-07 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2019-12

CONDITIONS: Neurodegenerative Diseases; Amyotrophic Lateral Sclerosis; Multiple Sclerosis; Parkinson Disease
Keywords: neurodegenerative diseases; amyotrophic lateral sclerosis; multiple sclerosis; Parkinson's Disease
MeSH Terms: conditions — Neurodegenerative Diseases; Amyotrophic Lateral Sclerosis; Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, feces
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subjects with ALS: subjects diagnosed with amyotrophic lateral sclerosis
- subjects with non-ALS neurodegenerative disease: subjects diagnosed with non-ALS neurodegenerative disease
- healthy controls: healthy subjects as controls

SUMMARY:
The etiology of many neurodegenerative diseases is unknown. A few studies have suggested the role of infection in the gastrointestinal tract in the etiology and pathogenesis of neurological diseases such as idiopathic Parkinson. For example, infection with Helicobacter pylori has been suggested to play a role in Parkinson disease. In addition, bacterial pathogens such as spirochetes and bacterial products such as cyanobacterial toxins have been speculated as the contributing factors in the development of amyotrophic lateral sclerosis (ALS). The effect of microbial composition of the gut in the pathogenesis of ALS is suspected. The difference in the bacterial profile of the gut has been documented in diseases such as inflammatory bowel disease and obesity.

The goal of this IRB protocol is to create a human tissue bank and to obtain patients' demographic information for future investigation of the role of bacterial pathogens and the role of gut flora composition in the development of neurodegenerative diseases including but not limited to ALS, Parkinson's disease, and multiple sclerosis.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to create a bank of fecal and blood samples and associated coded demographic information for future investigation of the microbial etiology and pathophysiology of neurodegenerative diseases including but not limited to Amyotrophic Lateral Sclerosis (ALS), Parkinson's disease and multiple sclerosis.

Approximately 300 adult participants (open to all races and both sexes) subjects will be recruited (i.e. 100 healthy controls, 100 subjects with other neurodegenerative diseases (not ALS) and 100 subjects with ALS).

Inclusion criteria permit all adults aged >18 years of age with the diagnosis of ALS who are willing to provide informed consent and patients who do not have a diagnosis of ALS and are willing to provide informed consent. Subjects who do not provide informed consent, have acute bacterial infection of the GI tract, and/or are being treated with antibiotics or probiotics within 28 days prior to sampling are excluded. A separate blood sample will not be taken from a subject if the maximum amount of samples allowed have been collected for standard care.

Upon arrival to the clinic, staff will provide the stool tissue bank protocol informed consent / HIPAA authorization document to eligible subjects for review. If subjects indicate a willingness to participate, the research coordinator or one of the participating investigators will review the informed consent form / HIPAA authorization with the subjects and answer any questions. If subjects agree to participate, they will sign the informed consent form / HIPAA authorization. Copies of the document will be made for subjects; originals will be filed in a locked cabinet.

Biological materials will be collected from the patient using either one or both of the following methods: as biological samples obtained specifically for the study (e.g. stool samples from all participating patients) or as extra material obtained specifically for research in addition to material collected as part of routine care (e.g., blood samples).

Subjects will be asked to consider participating in the stool tissue bank protocol. If subjects consent to donate extra samples for the bank, the samples will be obtained by the physicians or the clinic staff.

Two 10 ml venous blood samples for the ALS tissue bank will be collected 1) in a serum separator, and 2) in a tube containing the anticoagulant, EDTA (lavender top). Stool samples will be collected in sterile plastic cups. The blood and stool samples will be put on ice or refrigerated as promptly as possible until delivered to the ALS Research Laboratory at Cannon Research Center.

Samples will be de-identified by labeling with a research code prior to entering the laboratory. All information pertaining to the sample including a copy of the consent form and the master list of the research coding will be secured in a locked file cabinet. Personal health information (PHI) obtained will be entered into a separate security-protected database utilizing encryption technology and accessible only to authorized personnel. The samples, once coded, will be given to the appropriate laboratory technician for processing and analysis.

Blood samples will be centrifuged, the plasma and serum samples will be aliquoted in 1 ml tubes and stored at -80 C. The blood cells, separated from plasma, will be processed for DNA isolation immediately or stored at -80 C for later DNA extraction. Four ~25 mg aliquots of stool samples will be stored in sterile tubes at -80 C for future analysis. Storage freezers are locked, connected to emergency power and monitored by an alarm system that notifies laboratory personnel of malfunctions, etc.

In addition, a data collection form will be completed by the research staff to collect demographic, medical history, etc. as shown in Appendix C. The form will be linked to the tissue samples by an individual research code. This information is necessary for defining the tissue samples collected.

No formal sample size determination will be performed for this tissue bank protocol.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* patients diagnosed with amyotrophic lateral sclerosis or other neurodegenerative disease, and healthy controls

Exclusion Criteria:

* Subjects with acute bacterial infection of the GI tract
* Subjects on treatments with antibiotics or probiotics within 28 days prior to sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at Carolinas Medical Center with and without neurodegenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12-02 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Creation of a bank of fecal and blood samples to study the mirobial etiology of neurodegenerative diseases | one year
  The goal of this protocol is to create a human tissue bank of fecal and blood samples for the future investigation of the microbial etiology and pathophysiology of neurodegenerative diseases including but not limited to Amyotrophic Lateral Sclerosis, Parkinson's Disease, and Multiple Sclerosis. Patient demographic information will be collected to allow future study of the role of bacterial pathogens and gut flora composition in the development of neurodegenerative diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, MD, Principal Investigator — Director, Neuromuscular ALS/MDA Center and Neuromuscular/ALS Research Laboratory
Locations (1):
- Carolinas Medical Center - Dept of Neurology, Charlotte, North Carolina, United States